CLINICAL TRIAL: NCT01158625
Title: Nighttime Dosing of Antihypertensive Drugs in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Regionshospitalet Silkeborg (Other); The Ministry of Science, Technology and Innovation, Denmark (Other Government); Central Denmark Region (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: M-20100084
Record Dates: First submitted 2010-06-25; First posted 2010-07-08 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Diabetes Mellitus, Type 2; Hypertension
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Morning dosing of antihypertensive drugs (No Intervention)
- Nighttime dosing of antihypertensive drugs (Active Comparator)
  Interventions: Other: Change of time of administration

INTERVENTIONS:
Other: Change of time of administration — Change of time of administration
  Arms: Nighttime dosing of antihypertensive drugs

SUMMARY:
The purpose of this study is to investigate if it is possible to lower the nighttime blood pressure in patients with type 2 diabetes mellitus by shifting the administration of antihypertensive drugs from morning to nighttime.

DETAILED DESCRIPTION:
In recent years several studies have shown that high nighttime blood pressure is associated with increased cardiovascular risk independently of the average 24 hour blood pressure. As a consequence there has been increasing focus on nighttime blood pressure and how to lower it. One way of addressing the problem is to shift the administration of antihypertensive drugs from morning to nighttime. Studies on non-diabetic patients show that by doing this the nighttime blood pressure can be lowered with 3-5 mm Hg without negative effect on the 24 hour blood pressure.

Only recently a study was made on diabetic patients. This showed similar results as for non-diabetic patients.However this study was based on diabetic patients who did not receive any antihypertensive drugs before.

This study will investigate the effects on nighttime blood pressure when shifting administration of antihypertensive drugs from morning to nighttime. The population is diabetic patients who are already in antihypertensive treatment.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Systolic nighttime blood pressure above 120 mm Hg
* Systolic daytime blood pressure not exceeding 150 mm Hg
* Antihypertensive treatment which must include
* once-daily drugs
* at least one drug must be a Angiotensin-Converting Enzyme Inhibitor, Angiotensin II Receptor Blocker or Renin Inhibitor.

Exclusion Criteria:

* MI or stroke within 6 months
* heart failure (EF < 45 %)
* atrial fibrillation
* eGFR < 30 ml/min

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2010-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Blood pressure, nighttime blood pressure and 24 h blood pressure | After 16 weeks

SECONDARY OUTCOMES:
Urine albumin excretion | After 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Klavs W Hansen, MD, DrMedSc, Study Director — Department of Medicine, Regional Hospital Silkeborg
Locations (2):
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Regional Hospital Silkeborg, Silkeborg